CLINICAL TRIAL: NCT05657470
Title: Rescue Thrombolysis for Medium Vessel Occlusion (RESCUE-TNK): a Prospective, Randomized, Open-label, Blinded End Point, and Multicenter Trial
Brief Title: Rescue Thrombolysis for Medium Vessel Occlusion (RESCUE-TNK)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Collaborators: Cerebrovascular Disease Collaboration & Innovation Alliance of Liaoning (Unknown)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2022) 187
Record Dates: First submitted 2022-12-02; First posted 2022-12-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNK group (Experimental)
  Interventions: Drug: Tenecteplase
- control group (No Intervention)

INTERVENTIONS:
Drug: Tenecteplase — intra-arterial tenecteplase
  Arms: TNK group

SUMMARY:
The best reperfusion strategy for medium-sized vessel occlusion (MeVO) is not well established. Given the proven treatment effect of intra-arterial thrombolysis in patients with large vessel occlusion (LVO), the investigators hypothesized that intra-arterial tenecteplase (TNK) could increase the recanalization rate of MeVO and thus improve clinical outcome. The current study aimed to explore the safety and efficacy of intra-arterial TNK in patients with MeVO.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Medium vessel occlusion (MeVO), referring to M2-3 of MCA; A1-3 of ACA; P1-3 of PCA; PICA, AICA or SCA (including primary, distal embolism in the same region after thrombectomy or concurrent embolism in other regions).

   * Primary MeVO as detected by the first DSA examination or secondary MeVO after mechanical thrombectomy for large vessel occlusion;
   * MeVO causes neurological deficits in motor strength, language, vision etc;
   * Endovascular mechanical thrombectomy cannot be performed as assessed by the investigator;
   * Absence of parenchymal hematoma on CT images performed in the angio suite.
3. Within 24 hours from symptom onset;
4. Signed informed consent by patient or patient's legally authorized representative.

Exclusion Criteria:

1. Patients with completed infarction in the territory of the MeVO on non-contrast CT;
2. Patients with intracranial hemorrhage;
3. Coagulation disorders, tendency for systemic hemorrhagic, thrombocytopenia (<100,000/mm3);
4. Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
5. After mechanical thrombectomy, severe and sustained (> 5 minutes) uncontrolled hypertension (systolic blood pressure over 180mmHg or diastolic blood pressure over 105 mmHg);
6. Patients with contraindication or allergy to any ingredient of study medication;
7. Pregnancy, plan to get pregnant or active lactation;
8. The estimated life expectancy is less than 6 months due to other serious diseases;
9. Other conditions unsuitable for this clinical study as assessed by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
proportion of patients with successful Medium vessel occlusion (MeVO) recanalization | immediately after finishing intra-arterial tenecteplase
  successful MeVO recanalization is defined as the expanded treatment in cerebral ischemia (eTICI) score 2b67-3 in the territory of the target occluded MeVO artery

SECONDARY OUTCOMES:
proportion of modified Rankin Scale (mRS) 0-1 | Day 90
  mRS scores range from 0 to 6, with higher scores indicating worse outcome
proportion of modified Rankin Scale (mRS) 0-2 | Day 90
  mRS scores range from 0 to 6, with higher scores indicating worse outcome
distribution of modified Rankin Scale (mRS) | Day 90
  mRS scores range from 0 to 6, with higher scores indicating worse outcome
incidence of early neurological improvement | 24 (-6/+24) hours
  early neurological improvement is defined as a decrease of more than 4 points or reaching 0 points in NIHSS score, compared with baseline
Changes in National Institute of Health stroke scale (NIHSS) | 24 (-6/+24) hours
  NIHSS scores range 0-42, with higher scores indicating greater stroke severity
rate of visual recovery in patients with posterior cerebral artery occlusion | 7 days or at hospital discharge
proportion of symptomatic intracranial hemorrhage | 24 (-6/+24) hours
  symptomatic intracranial hemorrhage is defined as an increase in the NIHSS score of ≥4 points as a result of the intracranial hemorrhage
proportion of parenchymal hematoma type 1 and 2 | 24 (-6/+24) hours
all serious adverse events | 24 (-6/+24) hours
all-cause death | 7 days
recurrent stroke, cardiovascular events, other vascular events and death | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided